CLINICAL TRIAL: NCT06767020
Title: A Multi-center Comparative Real-World Study on AQP4 Antibody Detection Methods Using Live Cell and Fixed Cell-Based Assay Technologies
Brief Title: Comparative Study on AQP4 Antibody Detection Methods
Status: Active, not recruiting | Type: Observational
Sponsor: First Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Feng Jinzhou, Ph.D, First Affiliated Hospital of Chongqing Medical University
Other Study IDs: AQP4NMO-001
Record Dates: First submitted 2025-01-04; First posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: NMOSD
Keywords: AQP4; Fixed CBA; Live CBA

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 120 Days
Biospecimen Retention: Samples With DNA — Blood samples are collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- NMOSD: cases confirm a diagnosis of NMOSD according to 2015 NMOSD diagnostic criteria by IPND (International Panel for NMO Diagnosis).
- suspected NMOSD: cases having features suggestive of NMOSD but can not confirm a diagnosis of NMOSD according to 2015 NMOSD diagnostic criteria by IPND (International Panel for NMO Diagnosis).
- MS: cases confirm a diagnosis of MS according to 2017 McDonald criteria with no features suggestive of NMOSD.
- Other disease: cases confirm a diagnosis of neurological disease other than NMOSD and MS, including autoimmune encephalitis, viral encephalitis, myasthenia gravis et al.

SUMMARY:
This study aims to determine which method is more suitable for clinical application by comparing the sensitivity, specificity, and accuracy of serum AQP4-IgG detection using live cell CBA and fixed cell CBA methods, thereby improving the diagnostic accuracy of neuromyelitis optica spectrum disorders (NMOSD).

DETAILED DESCRIPTION:
This is a multi-center comparative real-world study on AQP4 Antibody Detection Methods Using Live Cell and Fixed Cell-Based Assay Technologies. This study aims to determine which method is more suitable for clinical application by comparing the sensitivity, specificity, and accuracy of serum AQP4-IgG detection using live cell CBA and fixed cell CBA methods, thereby improving the diagnostic accuracy of neuromyelitis optica spectrum disorders (NMOSD). One hundred and twenty patients from 3 centres in China will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* NMOSD: Confirm a diagnosis of NMOSD according to 2015 NMOSD diagnostic criteria by IPND (International Panel for NMO Diagnosis) suspected NMOSD: cases having features suggestive of NMOSD but can not confirm a diagnosis of NMOSD according to 2015 NMOSD diagnostic criteria by IPND (International Panel for NMO Diagnosis).

the following 'high risk' clinical and laboratory features had to be met

1. optic neuritis that was either severe with poor recovery (residual visual acuity in better eye worse or equal to 6/36), bilateral (simultaneous orsequential within 3 months) or recurrent (more than 2 attacks) as the sole clinical manifestation of demyelinating disease,
2. severe transverse myelitis with a central cord syndrome (symmetrical, motor, sensory and bladder involvement) and poor recovery (residual EDSS greater than 5.0) or a longitudinally extensive lesion of the spinal cord spanning 3 or more vertebral segments on magnetic resonance imaging (MRI) or
3. demyelinating disease clinically confined to the optic nerve and spinal cord with at least one of the following: normal or atypical MRI of the brain (fewer than 2 periventricular lesions), negative oligoclonal bands in cerebrospinal fluid, raised CSF protein or a CSF pleocytosis (more than 10 cells per μl) 2.All subjects provided written informed consent.

Exclusion Criteria:

* 1.Patients with incomplete clinical information. 2.Patients without serum samples.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Sex, Gender, diagnose, the number of relapses in NMOSD patients
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-11-11 (Actual); Primary Completion 2025-01-27 (Estimated); Study Completion 2025-01-27 (Estimated)

PRIMARY OUTCOMES:
Sensitivity (CI%), Specificity (CI%), Accuracy (CI%), PLR (CI%), NLR (CI%) | immediately
  The sensitivity, 95% confidence interval (CI) for sensitivity, specificity, and 95% CI for specificity of AQP4 antibody detection methods using live cell and fixed cell-based assay technologies in NMOSD and suspected NMOSD, along with the corresponding results from various control groups and overall controls, are given.

SECONDARY OUTCOMES:
Agreement ,Cohen's kappa, Spearman correlation coefficient | immediately
  The agreement ,Cohen's kappa, Spearman correlation coefficient of serum AQP4 antibody detection results using live CBA and fixed CBA.

CONTACTS AND LOCATIONS:
Overall Officials: Jinzhou Feng, Ph.D, Principal Investigator — First Affiliated Hospital of Chongqing Medical University
Locations (1):
- First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No